CLINICAL TRIAL: NCT05660642
Title: An Open-Label, Phase 2a Study to Evaluate the Safety, Tolerability and Pharmacodynamics of BPL-003 in Patients With Treatment Resistant Depression
Brief Title: An Open-Label Study to Evaluate the Safety, Tolerability and Pharmacodynamics of BPL-003 in Patients With Treatment Resistant Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-003-204
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: BPL-003
- Arm B (Experimental)
  Interventions: Drug: BPL-003

INTERVENTIONS:
Drug: BPL-003 — Experimental BPL-003 arms: will investigate one of two doses of BPL-003 (Part 1) and two doses of BPL-003 (Part 2)

SUMMARY:
An open-label, multi-centre, Phase 2a study to evaluate the safety, tolerability, and pharmacodynamics of one and two doses of intranasal BPL-003 combined with psychological support, in patients with treatment resistant depression when administered as monotherapy or as adjunctive therapy with defined SSRIs (citalopram, escitalopram, sertraline or fluoxetine).

DETAILED DESCRIPTION:
Part 1: Up to 32 patients, across 2 parallel arms (Arms A and Arms B) will receive one of two single doses of BPL-003, given intranasally, with 12 weeks of follow-up assessments.

Part 2: Up to 32 patients, across 2 parallel arms (Arms A and Arms B) will receive two doses of BPL-003, given intranasally, with 10 weeks of follow-up assessments.

Psychological support will be given before, during and after dosing in Part 1 and Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Major Depressive Disorder.
2. Diagnosed with TRD defined as failure to respond to an adequate dose and duration of at least 2 pharmacological treatments in the past 5 years prior to screening, at least one of which is during the current episode.
3. Montgomery-Asberg Depression Rating Scale score ≥24 at Screening.
4. Clinical Global Impression - Severity ≥4 at Screening.
5. Willing and able to discontinue current pharmacological anti-depressant therapy.
6. On current stable dose of pharmacological antidepressant therapy limited to one of 4 SSRIs (Arm B), i.e. either citalopram, escitalopram, sertraline or fluoxetine.

Exclusion Criteria:

1. Current or history of schizophrenia, psychotic disorder including psychotic depression, bipolar disorder, delusional disorder, schizoaffective disorder, or any other severe psychiatric disorder.
2. Current personality disorders.
3. First-degree family history of schizophrenia, bipolar disorder, delusional disorder, personality disorders or schizoaffective disorder.
4. Current alcohol or substance use disorder (other than caffeine or nicotine).
5. A participant who at any time, has been unresponsive to ketamine, esketamine, an adequate course of treatment with electroconvulsive therapy, or has received vagal nerve stimulation or deep brain stimulation.
6. Suicidal ideation with the intent to act or suicidal behaviour within the 12 months prior to the start of Screening or on Day 1 prior to dosing.
7. Suicide attempt and/or self-injurious behaviour within the last 12 months prior to Screening.
8. Uncontrolled medical conditions e.g. hypo/hyperthyroidism, diabetes, renal failure.
9. Seizure disorder or history of seizures (including febrile seizures).
10. Abnormal and clinically significant results on the physical examination, vital signs, electrocardiogram, or laboratory tests at Screening Baseline.
11. Any nasal obstruction, blockage, or symptoms of congestion at the time of dosing, that in the Investigator's opinion may interfere with administration of the study drug.
12. Currently receiving lithium, antipsychotics, serotonergic drugs (excluding the permitted SSRIs for arm B), psychostimulants, or any other prohibited medication.
13. Female patients who are pregnant or lactating, or of childbearing potential and not willing to use adequate forms of contraception.
14. Male patients who are sexually active and not willing to using adequate forms of contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
1. To assess the safety and tolerability of single or multiple intranasal doses of BPL-003 in patients with treatment resistant depression | Baseline to 12 weeks post dose
  * Percentage of patients with treatment emergent adverse events
  * Percentage of patients with clinically significant abnormal laboratory tests
  * Percentage of patients with clinically significant abnormal vital signs
  * Percentage of patients with clinically significant findings in physical examination
  * Percentage of patients with clinically significant ECG parameters or cardiac telemetry abnormalities (Part 1 Arm B only)
  * Percentage of patients with suicidal ideation or behaviour

OTHER OUTCOMES:
Change from Baseline in MADRS | Day 2 to 12 weeks post dose
Percentage of responders | Day 2 to 12 weeks post dose
  Defined as 50% reduction in MADRS score compared to Baseline
Percentage of patients in remission | Day 2 to 12 weeks post dose
  Defined as MADRS score of <11
Plasma levels of 5-MeO-DMT and its metabolites | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: VP and Head of Clinical Development, PhD, Study Director — Beckley Psytech Ltd
Locations (3):
- United Kingdom (3):
  - MAC Clinical Research, Liverpool
  - Hammersmith Medicines Research, London
  - King's College London, Clinical Trials Facility, London

IPD SHARING:
Plan to Share IPD: No
Due to the UK GDPR, individual participant data will not be shared publicly. Group data will be presented in publication after study completion.